CLINICAL TRIAL: NCT02388763
Title: Clinical Evaluation of MyDay™ Daily Disposable Silicone Hydrogel Contact Lenses
Brief Title: Clinical Evaluation of MyDay™ and 1-DAY ACUVUE® TruEye®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CLY838-P001
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Refractive Error
Keywords: Contact lenses
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MyDay, then 1DAVTE (Other): Stenfilcon A contact lenses, followed by narafilcon A contact lenses. Each product worn bilaterally (in both eyes) for 10 days in a daily wear, daily disposable modality.
  Interventions: Device: Stenfilcon A contact lenses; Device: Narafilcon A contact lenses
- 1DAVTE, then MyDay (Other): Narafilcon A contact lenses, followed by stenfilcon A contact lenses. Each product worn bilaterally for 10 days in a daily wear, daily disposable modality.
  Interventions: Device: Stenfilcon A contact lenses; Device: Narafilcon A contact lenses

INTERVENTIONS:
Device: Stenfilcon A contact lenses — Contact lenses worn during Period 1 or 2, as randomized
  Other Names: MyDay™
Device: Narafilcon A contact lenses — Contact lenses worn during Period 1 or 2, as randomized
  Other Names: 1-DAY ACUVUE® TruEye®

SUMMARY:
The purpose of this study is to evaluate the functional vision of 2 daily disposable silicone hydrogel contact lenses using Time Controlled Visual Acuity (TCVA) measurements at high luminance and high contrast after 10+/-3 days of wear post 3 hour exposure to a reduced humidity environment.

DETAILED DESCRIPTION:
After randomization, participants attended a baseline visit to include a 3 hour exposure to reduced humidity environment. The participant's habitual lenses were worn for the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Must sign informed consent form.
* Adapted, current soft silicone hydrogel daily disposable contact lens wearer during the last 2 months.
* Willing to wear lenses every day or at least 5 days per week 6 hours per day.
* Willing to discontinue artificial tears and rewetting drops usage on the days of study visits.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Monocular (only 1 eye with functional vision) or fit with only 1 lens.
* Pregnant or lactating.
* Current MyDay™ or 1DAY ACUVUE® TruEye® lens wearer.
* Any abnormal ocular condition as specified in the protocol.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Manager, EMEA, Study Director — Alcon, A Novartis Division

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 1 investigative site located in the United Kingdom.
Pre-assignment Details: Of the 66 enrolled participants, 2 participants were discontinued prior to randomization. This reporting group includes all randomized participants (64).
Groups:
- Habitual, MyDay, 1DAVTE: Habitual contact lenses worn first, followed by stenfilcon A contact lenses in Period 1 and narafilcon A contact lenses in Period 2. Each product worn bilaterally for 10 days in a daily wear, daily disposable modality.
- Habitual, 1DAVTE, MyDay: Habitual contact lenses worn first, followed by narafilcon A contact lenses in Period 1 and stenfilcon A contact lenses in Period 2. Each product worn bilaterally for 10 days in a daily wear, daily disposable modality.
Period: Habitual, 10 Days of Wear
Arm/Group | Habitual, MyDay, 1DAVTE | Habitual, 1DAVTE, MyDay
Started | 32 | 32
Completed | 31 | 31
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Period 1, 10 Days of Wear
Arm/Group | Habitual, MyDay, 1DAVTE | Habitual, 1DAVTE, MyDay
Started | 31 | 31
Completed | 30 | 30
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Period 2, 10 Days of Wear
Arm/Group | Habitual, MyDay, 1DAVTE | Habitual, 1DAVTE, MyDay
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This reporting group includes all randomized participants.
Groups:
- Overall: Habitual contact lenses worn first, followed by stenfilcon A contact lenses and narafilcon A contact lenses in Periods 1 and 2 as randomized. Each product worn bilaterally for 10 days in a daily wear, daily disposable modality.
Arm/Group | Overall
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: High Contrast Time-Controlled Visual Acuity (TCVA) (VA Unit) Post-Exposure to Reduced Humidity at Day 10
Description: High contrast TCVA was assessed after 3 hours exposure to reduced humidity environment. TCVA test was performed at 4 meters under high illumination (90%) using a Landolt ring test. For each acuity level, a series of single rings with gaps in one of four directions was presented and the percentage of correctly identified rings constituted the score. TCVA was measured in VA units and a higher TCVA value indicates an improvement in visual acuity. Both eyes contributed to the analysis.
Time Frame: Day 10, each product
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: VA unit
Groups:
- MyDay: Stenfilcon A contact lenses worn bilaterally for 10 days in a daily wear, daily disposable modality
- 1DAVTE: Narafilcon A contact lenses worn bilaterally for 10 days in a daily wear, daily disposable modality
Arm/Group | MyDay | 1DAVTE
Number analyzed (Participants) | 60 | 60
VA unit | 0.453 (0.673) | 0.341 (0.781)

2. Secondary Outcome: High Contrast TCVA (VA Unit) Pre-Exposure to Reduced Humidity at Day 10
Description: High contrast TCVA was assessed after 3 hours exposure to normal environment and prior to exposure to reduced humidity environment. Both eyes contributed to the analysis.
Time Frame: Day 10, each product
Population: Intent to Treat Subjects
Measure: Mean (Standard Deviation); unit: VA unit
Arm/Group | MyDay | 1DAVTE
Number analyzed (Participants) | 60 | 60
VA unit | 0.614 (0.689) | 0.700 (0.777)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of informed consent throughout the duration of a subject's participation in the study (up to 30 days). This analysis population includes all randomized participants exposed to investigational product (habitual, MyDay, and 1DAVTE) from time of product dispense (safety analysis set), based on treatment-specific exposure. One subject in the MyDay/1DAVTE arm wore habitual lenses during Period 1 and was not exposed to MyDay (discontinued at Period 1).
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the medical device. Ocular AEs are presented on the subject level, but reported by eye.
Groups:
- Pretreatment: All subjects who consented to participate in the study prior to the initiation of study treatment
- Dailies Total 1: Delefilcon A contact lenses per subject's habitual prescription worn for 10 days prior to Period 1
- Clariti 1-Day: Somofilcon A contact lenses per subject's habitual prescription worn for 10 days prior to Period 1
- MyDay: Stenfilcon A contact lenses worn for 10 days during Period 1 or 2 as randomized
- 1DAVTE: Narafilcon A contact lenses worn for 10 days during Period 1 or 2 as randomized
Arm/Group | Pretreatment | Dailies Total 1 | Clariti 1-Day | MyDay | 1DAVTE
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/32 | 0/32 | 1/60 | 1/61
Other Adverse Events (participants affected / at risk) | 0/66 | 5/32 | 0/32 | 0/60 | 0/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=66) | Dailies Total 1 (N=32) | Clariti 1-Day (N=32) | MyDay (N=60) | 1DAVTE (N=61)
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Renal vein thrombosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=66) | Dailies Total 1 (N=32) | Clariti 1-Day (N=32) | MyDay (N=60) | 1DAVTE (N=61)
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 2 | 0 | 0 | 0 — Incidences of hordeolum occurred in 2 out of 64 eyes (3.1%), here reported as 2/32 (6.25%) in order to keep all AE reports on the subject level.
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 — Incidences of foreign body in eye occurred in 2 out of 64 eyes (3.1%), here reported as 2/32 (6.25%) in order to keep all AE reports on the subject level.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.